CLINICAL TRIAL: NCT01793818
Title: Evaluation on Seropositive Patients of a Synthetic Vaccine Targeting the HIV Tat Protein
Acronym: EVATAT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BIOSANTECH (Industry)
Collaborators: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EVATAT
Record Dates: First submitted 2013-02-14; First posted 2013-02-18 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: AIDS
Keywords: Vaccine; HIV-1; Tat
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 Phase I/II (Placebo Comparator): Three injections with no active principle
  Interventions: Biological: Tat Oyi
- Group 2 Phase I/II (Active Comparator): Three injections of Tat Oyi vaccine containing 11 µg of active principle
  Interventions: Biological: Tat Oyi
- Group 3 Phase I/II (Active Comparator): Three injections Tat Oyi vaccine containing 33 µg of active principle
  Interventions: Biological: Tat Oyi
- Group 4 Phase I/II (Active Comparator): Three injections Tat Oyi vaccine containing 99 µg of active principle
  Interventions: Biological: Tat Oyi

INTERVENTIONS:
Biological: Tat Oyi — Three injections in the arm

SUMMARY:
Tat Oyi vaccination on seropositive patients could help their immune system to recognize and neutralize Tat. The neutralization of extra cellular Tat should help the cellular immune response to eliminate HIV-1 infected cells.

DETAILED DESCRIPTION:
The protocol got a favorable judgment from an ethic committee (CPP SudMed 2) on November 9th, 2012 and was authorized by the French drug agency (ANSM) on January 24th, 2013. It will be proposed to HIV-1 infected volunteers to participate to a phase I/II clinical trial to test the Tat Oyi vaccine. Volunteers will have an undetectable viremia (lower than 40 copies/ml) and a level of CD4 cells higher than 350 /mm3 since at least one year under Anti Retroviral Treatment (ART). It will be a randomized double blinded clinical trial with a placebo.

Main Objective: No undesirable events due to vaccination and viremia remaining < 100 copies/ml after interruption of cART.

Secondary objective: An immune response against Tat characterized by the cross recognition of Tat variants representative of the five main HIV-1 clades.

Main parameter of evaluation: Plasma viremia. Secondary parameter of evaluation: Detection with ELISA of antibodies able to recognize Tat variants representative of the five main HIV-1 clades.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 64 years old for the pre inclusion visit.
* Documented HIV-1 Infection
* Preferentially, group A patients from CDC classification but no group C patients.
* HIV-1 patients treated with three antiretroviral drugs since 12 months not changed since three months and having an undetectable viremia since 12 months.
* HIV-1 Chronic infection defined by a positive HIV-1 ELISA and HIV-1 proteins characterized in a full HIV-1 Western blot. Stable undetectable plasmatic HIV RNA (lower than 40 copies/ml) since 12 months. Lymphocyte CD4 cells higher than 350/mm3 with a NADIR higher than 200/mm3 since 12 months.
* Free engagement, fully explained and wrote with the patient signature for the inclusion visit and before any test required for the clinical trial.
* Patient affiliated to a social security system.
* No vaccination against influenza or other pathogens since three months.
* No chemotherapy or treatments with corticosteroid
* HIV-1 patients being abstinent former drug users or drug users following substitution training.

Exclusion Criteria:

* HIV-1 patient protected regarding French law (articles L1121-5, L1121-6, L1121-7, L1121-8 & L1122-2)
* No HIV-1 infection
* Patient infected with HIV-2
* Patient in HIV-1 primo infection or recently in primo infection
* Patient in symptomatic primo infection or CD4 cells lower than 200/mm3
* Women sexually active with no efficient contraception
* Pregnant women or brass feeding.
* Patient with an opportunistic infection in the CDC group C.
* Patient with a cancer and/or under chemotherapy or radiotherapy.
* Patient with an evolutive psychiatric pathology
* Patient being HBV and/or HCV positive
* Patient being ELISA positive for HTLV-1
* Patient being cirrhotic (Child and Pugh level A, B and C)
* Patient under criminal investigation
* Patients with abnormal blood formulation
* Patient participating to another clinical research

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-02; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Optimal vaccine dose (phase I/II) | Two years
  No undesirable events due to vaccination and viremia remaining < 100 copies/ml after interruption of ART.

SECONDARY OUTCOMES:
Optimal Vaccine Dose (phase I/II) | Two years
  An immune response against Tat characterized by the cross recognition of Tat variants representative of the five main HIV-1 clades.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Ravaux, MD, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Centre d'Investigation Clinique - Universitary Hospital Centre Conception, Marseille, France

IPD SHARING:
Plan to Share IPD: Yes
Data base (HIV RNA, CD4, CD8, HIV DNA, Tat immune response) and statistical analysis

REFERENCES:
- [Background] Loret E. HIV extracellular Tat: myth or reality? Curr HIV Res. 2015;13(2):90-7. doi: 10.2174/1570162x12666141202125643. PMID 25439235